CLINICAL TRIAL: NCT02742363
Title: Long Term Oral and Dental Effects in Adolescents Who Were Treated for Cancer in Childhood
Brief Title: Long Term Dental Effects in Adolescents Who Were Treated for Cancer in Childhood
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: 0004-16-HMO-CTIL
Record Dates: First submitted 2016-03-23; First posted 2016-04-19 (Estimated); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Other: Collecting data — Collecting data from patient records

SUMMARY:
The investigators aim is to explore associations between specific types of cancer therapy, age at treatment and the presence of dental abnormalities in adolescence.

The study will help identify unique dental changes, malformations and or missing teeth that appear in adolescence as a secondary complication due to anticancer treatment (chemotherapy and or radiotherapy) given in childhood.

Materials and methods:

* Study Group: 200 patients, at least 12 years old, who were treated for Cancer at the age of 0-10 years old.
* The following data will be collected: Demographic information, Medical Status, Cancer therapy, Intraoral examination, Oral soft and hard tissue condition and radiographic examination.

ELIGIBILITY:
Inclusion Criteria:

* were treated for Cancer at the age of 0-10 years old

Exclusion Criteria:

* None

Ages: 12 Years to 32 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients, at least 12 years old, who were treated for Cancer at the age of 0-10 years old. The maximum time span of entering the study group-up to 20 years after last session of oncology treatment.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Oral abnormalities associated with cancer therapy. | Two years
  A medical survey will be filled out with the patient and his legal guardian. A full dental examination will gather all clinical and radiographic findings. The following measures will be noted:
  1. Description of chemotherapy agents and duration
  2. Radiotherapy continuation.
  3. Radiotherapy dosage in Gray units.
  4. Yes/No questions regarding previous dental trauma.
  5. Yes/No questions regarding previous dental treatment.
  6. Questions regarding oral hygiene.
  7. Questions concerning oral habits.
  8. Extra oral examination.
  9. Intra oral clinical findings will be listed by tooth number.
  10. Radiographic findings will be listed by tooth number.

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel